CLINICAL TRIAL: NCT03607812
Title: ABPM (Automatic Measurement of Blood Pressure) Evaluation in the Diagnosis and Management of Arterial Hypertension for Algerian Patients in Current Medical Practice
Brief Title: Diagnosis and Management of Arterial Hypertension for Algerian Patients in Current Medical Practice
Acronym: MAPADZ
Status: Completed | Type: Observational
Sponsor: Merinal Laboratoires (Industry)
Collaborators: Axelys Sante Dz (Industry)
Responsible Party: Sponsor
Other Study IDs: ASDZ_Obs_01_2017
Record Dates: First submitted 2018-05-09; First posted 2018-07-31 (Actual); Last update posted 2019-08-20 (Actual); Status verified 2019-08

CONDITIONS: Arterial Hypertension
Keywords: Hypertension; ABPM
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Blood pressure reduction and control are associated with reduced risk of stroke and cardiovascular disease. There is evidence that ambulatory blood pressure monitoring (ABPM) results more accurately reflect the risk of cardiovascular events than do office measurements of blood pressure. New international guidelines recognize the importance of ABPM which has an important and growing role in the diagnosis and in guiding antihypertensive therapy. In 2011 in the United Kingdom, the National Institute for Health and Care Excellence (NICE) recommended that ABPM be performed on all patients with suspected hypertension to confirm the diagnosis and reduce unnecessary treatment in people who do not have true hypertension. The aim of this observational study is to describe the utility of ABPM generally and specifically in the management of hypertension by Cardiologists in the Algerian context.

DETAILED DESCRIPTION:
The primary Objective of this study is to assess the benefit of the ABPM in the diagnosis and management of arterial hypertension in by Cardiologists.

The Secondary Objectives are:

* To identify the conditions of usage of ABPM for the diagnosis of arterial hypertension,
* To evaluate the blood pressure during the ABPM assessment and at 6 weeks of follow up
* To describe the study population (socio-demography),
* To describe the therapeutic stratégies and the compliance to treatment.

ELIGIBILITY:
Inclusion Criteria:

* Patients who are either hypertensive (defined as those with a clinic SBP ≥ 140 mmHg or DBP ≥ 90 mmHg [7]) or referred for the assessment of hypertension
* Informed consent obtained before any study-related activity

Exclusion Criteria:

* ABPM contraindication
* Patient with psychiatric disorder
* Patient not able to comply with study-related procedures based on clinical judgement of the investigator

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: In this observational study the target population will be constituted of patients who can benefit from the contribution of ABPM to confirm or refute (white coat effect) hypertension.
Sampling Method: Probability Sample
Enrollment: 1027 (Actual)
Dates: Start 2017-06-28 (Actual); Primary Completion 2018-07-31 (Actual); Study Completion 2018-08-31 (Actual)

PRIMARY OUTCOMES:
Diagnosis of hypertension | At 24 hours after the inclusion in the study (Visit 2)
  Valid 24h-ABPM: blood pressure ≥ 140/90 mmHg

SECONDARY OUTCOMES:
Patient Demography | At the Inclusion in the study
  Age, Sexe
Therapeutic Decison | At 24 hours after the inclusion in the study (Visit 2)
  * Initiation of antihypertensive therapy in naive patients if the dianosis of hypertension is confirmed.
  * Maintain, switch or adaptation of treatment in treated patients.
Self-measurement of Arterial blood Pressure | At 6 weeks after the inclusion in the study (Visit 3)
  Measurement of arterial pressure performed by the patient and reported on a follow up diary. Both systolic and diastolic pressures will be collected.
Evaluation of Compliance to treatment | At 6 weeks after the inclusion in the study (Visit 3)
  Evaluation test based on the method developed by Xavier Girerd, consisting in 6 questions on the compliance. The rating is divised in three categories: Good compliant, moderate compliant or non compliant. according to Girerd et al. Evaluation de l'observance par l'interrogatoire au cours du suivi des hypertendus dans des consultations spécialisées - Arch Mal Cœur Vaiss. 2001 Aug. 94-(8):839-42.

CONTACTS AND LOCATIONS:
Locations (1):
- Service de cardiologie EHS Maouche ( ex CNMS de Benaknoun), Algiers, Algeria

REFERENCES:
- [Background] Nansseu JR, Noubiap JJ, Mengnjo MK, Aminde LN, Essouma M, Jingi AM, Bigna JJ. The highly neglected burden of resistant hypertension in Africa: a systematic review and meta-analysis. BMJ Open. 2016 Sep 20;6(9):e011452. doi: 10.1136/bmjopen-2016-011452. PMID 27650760
- [Background] Nibouche WN, Biad A. [Arterial hypertension at the time of diagnosis of type 2 diabetes in adults]. Ann Cardiol Angeiol (Paris). 2016 Jun;65(3):152-8. doi: 10.1016/j.ancard.2016.04.017. Epub 2016 May 24. French. PMID 27234335
- [Background] Amrani A, Baba Hamed MB, Mesli Talebbendiab F. Association study between some renin-angiotensin system gene variants and essential hypertension in a sample of Algerian population: case control study. Ann Biol Clin (Paris). 2015 Sep-Oct;73(5):557-63. doi: 10.1684/abc.2015.1069. PMID 26489814
- [Background] Ghembaza MA, Senoussaoui Y, Tani MK, Meguenni K. Impact of patient knowledge of hypertension complications on adherence to antihypertensive therapy. Curr Hypertens Rev. 2014;10(1):41-8. doi: 10.2174/157340211001141111160653. PMID 25392143
- [Background] Lardjam-Hetraf SA, Mediene-Benchekor S, Ouhaibi-Djellouli H, Meroufel DN, Boulenouar H, Hermant X, Hamani-Medjaoui I, Saidi-Mehtar N, Amouyel P, Houti L, Goumidi L, Meirhaeghe A. Effects of established blood pressure loci on blood pressure values and hypertension risk in an Algerian population sample. J Hum Hypertens. 2015 May;29(5):296-302. doi: 10.1038/jhh.2014.81. Epub 2014 Sep 18. PMID 25231511
- [Background] Bachir Cherif A, Temmar M, Labat C, Atif L, Chibane A, Benkhedda S, Taleb A, Benfenatki N, Benetos A, Bouafia MT. [Cardiovascular morbimortality after a follow-up of six years in black hypertensive in South Algeria]. Ann Cardiol Angeiol (Paris). 2014 Jun;63(3):168-75. doi: 10.1016/j.ancard.2014.04.019. Epub 2014 May 15. French. PMID 24933716
- [Derived] Hammoudi-Bendib N, Manamani L, Ouabdesselam S, Ouamer DS, Ghemri S, Courouve L, Cherif A, Mahi L, Benkhedda S. Ambulatory Blood Pressure Monitoring in the Diagnosis and Management of Arterial Hypertension in Current Medical Practice in Algeria. Curr Hypertens Rev. 2021;17(1):75-82. doi: 10.2174/1573402116666200324144223. PMID 32208121